CLINICAL TRIAL: NCT02637921
Title: Planetary Habitat Simulation: The Combined Effects of Bed Rest and Normobaric Hypoxia Upon Bone and Mineral Metabolism (WP3)
Brief Title: Planetary Habitat Simulation: Bone Metabolism Studies
Acronym: PlanHab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Jozef Stefan Institute (Other); DLR German Aerospace Center (Other); KTH Royal Institute of Technology (Other); European Commission (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Dr, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 284438/WP3
Record Dates: First submitted 2015-12-01; First posted 2015-12-22 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Hypoxia; Bone Resorption
Keywords: bed rest; bone metabolism
MeSH Terms: conditions — Hypoxia; Bone Resorption | interventions — Ambulatory Care Facilities; Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hypoxic ambulatory (Active Comparator): Participants ambulatory in normobaric hypoxia with standardised nutritional intake
  Interventions: Other: Hypoxia; Other: Ambulatory; Other: Standardised nutritional intake
- Hypoxic Bed rest (Experimental): Participants are on bed rest in normobaric hypoxia with standardised nutritional intake
  Interventions: Other: Hypoxia; Other: Bed Rest; Other: Standardised nutritional intake
- Normoxic bed rest (Active Comparator): Participants are on bed rest in normobaric normoxia with standardised nutritional intake
  Interventions: Other: Normoxia; Other: Bed Rest; Other: Standardised nutritional intake

INTERVENTIONS:
Other: Hypoxia — 21 days confinement in normobaric hypoxic (FiO2 = 14%)
  Arms: Hypoxic Bed rest; Hypoxic ambulatory
Other: Ambulatory — Participants hava a standardized activity level throughout the intervention
  Arms: Hypoxic ambulatory
Other: Normoxia — 21 days confinement in normobaric normoxic (FiO2 = 21%) environment
  Arms: Normoxic bed rest
Other: Bed Rest — Participants remain on supine bed rest throughout the intervention
  Arms: Hypoxic Bed rest; Normoxic bed rest
Other: Standardised nutritional intake — Macronutrient, salt and dietary energy intake will be standardized per kg body weight for each participant

SUMMARY:
Bone losses are well known to occur in response to unloading (in microgravity or during immobilisation) and in patients with chronic obstructive airway disease (COPD). However, it is unknown whether there is an interactive effect between hypoxia and musculoskeletal unloading upon bone and mineral metabolism. Fourteen non-obese men, who are otherwise healthy, will undergo 3x 21-day interventions; normobaric normoxic bed rest (NBR; FiO2=21%), normobaric hypoxic ambulatory confinement (HAMB; FiO2=14%; ~4000 m simulated altitude), and normobaric hypoxic bed rest (HBR; FiO2=14%). The effects of hypoxia and bedrest on bone metabolism and phosphor-calcic homeostasis will be assessed (before and during each intervention, and 14 days after each intervention period) using venous blood sampling, 24hr urine collections, and peripheral quantitative computerized tomography (pQCT).

DETAILED DESCRIPTION:
The risk of bone loss in response to immobilization and space flight is widely recognized, with such bone losses occurring predominantly in the legs. Loading forces in the lower extremities are typically low in space and during bed rest, but musculoskeletal loading countermeasures can prevent or reduce bone losses induced in these conditions. Although the primary origin may be of a mechanical nature, bone losses in astronauts and immobilized patients are likely to be modulated by the endocrine and the internal environment.

Bone loss and osteoporosis is also prevalent in those with chronic obstructive pulmonary disease (COPD). The most discussed etiological factors for this condition include lack of physical activity, vitamin-D deficiency, hypogonadism, use of corticosteroids and smoking. However, COPD is associated with tissue hypoxemia and it is unclear whether hypoxia per se will affect bone turnover or metabolism.

The protocol of the current study standardises potential confounding factors, such as physical activity, ambient temperature, hypoxic stimulus and nutritional composition of the diet across all 3 interventions, and aims to extend our knowledge of the effects of hypoxia and bedrest on bone metabolism and phospho-calcic homeostasis.

Fourteen non-obese men, who are otherwise healthy, will be recruited following medical and psychological screening. They will be invited to attend the Olympic Sport Centre, Planica, Slovenia on 3 occasions, with each visit being 31 days in duration and separated by 5 months. Each 31-day visit ('campaign') includes a baseline recording period (5 days), 21 days of intervention, and a recovery period (5 days), with a follow-up visit being carried out 14 days after each intervention. The 3 interventions will be allocated in a randomized, cross over design: i) Normobaric normoxic bed rest (NBR; FiO2=21%), ii) Normobaric hypoxic ambulatory confinement (HAMB; FiO2=14%; ~4000 m simulated altitude), and iii) Normobaric hypoxic bed rest (HBR; FiO2=14%). A standardized, repeating, 14-day dietary menu, comprised of foods commonly consumed in the Slovenian diet, will be applied during all campaigns. Targeted energy intakes will be calculated individually using a modified Benedict-Harris formula, with physical activity factor multipliers of 1.2 for the HBR and NBR campaigns and 1.4 for the HAMB campaign, used to promote energy balance. Body mass will be monitored daily during the campaigns using a gurney incorporating load cells, and whole body composition will be determined before and immediately after each intervention using fan beam dual-emission X-ray absorptiometry. Macronutrient composition of the diet will be approximately 17% protein, 53% carbohydrate and 30% fat, with >1.1g of protein per kg body weight provided per day, and daily salt (sodium chloride) intake being <10g. Food will be provided in weighed portions and subjects will be encouraged to eat all food supplied. However, any food not eaten will be weighed and actual amount consumed recorded in a diet analysis programme.

Participants will have bone mineral content assessed at 5 time points (before, 3 during and one after each intervention) using pQCT scans of the calf and thigh. Horizontal scans will be taken at 4%, 14%, 38%, and 66% of the tibia (assessed from its distal end), and at 4% and 33% of the femur. Twenty-four hour urine collections will be obtained before (2 time points), during (11 time points) and after (3 time points) each intervention, and will be assessed for urinary calcium and phosphate content, and for a marker of bone reabsorption (N-terminal telopeptide). In addition, early morning, fasting venous blood samples will also be taken before (2 time points), and during (5 time points) each intervention. These will be analysed for calcium, phosphate, bone specific alkaline phosphatase, parathyroid hormone, 25-Hydroxyvitamin D, Procollagen-I-N-terminal propeptide and regulators of bone metabolism, (Dickkopf-related protein 1 and Sclerostin).

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy subjects
* Body mass index < 25 kg/m2
* Height 158 - 190 cm
* Waist circumference < 94 cm
* Volunteers that are able to declare their willingness to participate in the entire study
* Willing to be assigned randomly to the three groups
* Successfully passing the psychological and medical screening
* competent to sign informed consent
* Slovenian social insurance
* English language fluency

Exclusion Criteria:

* Medication required that may interfere with the interpretation of the results
* Bone mineral density (as measured by DEXA) more than 1.5 standard deviations < t score
* Recent sub-standard nutritional status
* Family history of thrombosis or positive response in thrombosis screening procedure.

(Biochemical analysis of the following parameters: ATIII, High sensitive C-reactive protein, S-Akt., Factor V-Leiden, Prothrombin, Lupus-partial thromboplastin time, Factor II)

* History of: thyroid dysfunction, renal stones, diabetes, allergies, hypertension, hypocalcemia, uric acidaemia, lipidaemia, or hyperhomocysteinaemia
* Gastro-esophageal reflux disease or renal function disorder, Hiatus hernia
* History of medical illness
* Smoker within six months prior to the start of the study
* Abuse of drugs, medicine or alcohol
* Participation in another study up to two months before study onset
* No signed consent form before the onset of the experiment
* Blood donors in the past three months before the onset of the experiment
* Vegetarian and Vegans
* Migraines
* History of orthostatic intolerance
* History of vestibular disorders
* Claustrophobia
* metallic implants, osteosynthesis material
* Chronic back pain

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral content, from baseline | 40 days
  assessed before (day -5), on days 2, 10 and 21 of the intervention and at the 14-day follow-up visit (40 days after 1st measurement) using pQCT scans of the calf and thigh.

SECONDARY OUTCOMES:
Change in urinary calcium concentration, from baseline | 30 days
  assessed from 24hr urine collections taken before (day -5), on days 1,2,3,4,8,10,12,14,16,18, and 21 of the intervention and on the 2nd, 3rd, and 4th day after each intervention period (last urine collection 30 days after first measurement)
Change in urinary phosphate concentration, from baseline | 31 days
  assessed from 24hr urine collections taken before (day -5), on days 1,2,3,4,8,10,12,14,16,18, and 21 of the intervention and on the 2nd, 3rd, and 4th day after each intervention period (last urine collection 31 days after first measurement)
Change in urinary N-terminal telopeptide concentration, from baseline | 31 days
  assessed from 24hr urine collections taken before (day -5), on days 1,2,3,4,8,10,12,14,16,18, and 21 of the intervention and on the 2nd, 3rd, and 4th day after each intervention period (last urine collection 31 days after first measurement)
Change in fasting serum calcium concentration, from baseline | 26 days
  assessed from venous blood samples taken before (day -5), and on days 2,5,10,14 and 21 of each intervention. Last sample point made 26 days after baseline sample
Change in fasting serum phosphate concentration, from baseline | 26 days
  assessed from venous blood samples taken before (day -5), and on days 2,5,10,14 and 21 of each intervention. Last sample point made 26 days after baseline sample
Change in fasting serum bone specific alkaline phosphatase concentration, from baseline | 26 days
  assessed from venous blood samples taken before (day -5), and on days 2,5,10,14 and 21 of each intervention. Last sample point made 26 days after baseline sample
Change in fasting serum parathyroid hormone concentration, from baseline | 26 days
  assessed from venous blood samples taken before (day -5), and on days 2,5,10,14 and 21 of each intervention. Last sample point made 26 days after baseline sample
Change in fasting serum 25-Hydroxyvitamin D concentration, from baseline | 26 days
  assessed from venous blood samples taken before (day -5), and on days 2,5,10,14 and 21 of each intervention. Last sample point made 26 days after baseline sample
Change in fasting serum Procollagen-I-N-terminal propeptide concentration, from baseline | 26 days
  assessed from venous blood samples taken before (day -5), and on days 2,5,10,14 and 21 of each intervention. Last sample point made 26 days after baseline sample
Change in fasting serum Dickkopf-related protein 1 concentration, from baseline | 26 days
  assessed from venous blood samples taken before (day -5), and on days 2,5,10,14 and 21 of each intervention. Last sample point made 26 days after baseline sample
Change in fasting serum Sclerostin concentration, from baseline | 26 days
  assessed from venous blood samples taken before (day -5), and on days 2,5,10,14 and 21 of each intervention. Last sample point made 26 days after baseline sample

CONTACTS AND LOCATIONS:
Overall Officials: Igor Mekjavic, PhD, Study Director — Jozef Stefan Institute; Jörn Rittweger, MD, PhD, Principal Investigator — German Aerospace Center (DLR)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rittweger J, Debevec T, Frings-Meuthen P, Lau P, Mittag U, Ganse B, Ferstl PG, Simpson EJ, Macdonald IA, Eiken O, Mekjavic IB. On the combined effects of normobaric hypoxia and bed rest upon bone and mineral metabolism: Results from the PlanHab study. Bone. 2016 Oct;91:130-8. doi: 10.1016/j.bone.2016.07.013. Epub 2016 Jul 18. PMID 27443510